CLINICAL TRIAL: NCT02605226
Title: A Prospective Multi-center Study to Compare the QOL and Efficacy of External Beam Radiation Therapy or Cryoablation Therapy for Stage III Prostate Cancer
Brief Title: Cryoablation Therapy or Radiotherapy Therapy for Stage III Prostate Cancer
Acronym: CRYO-PCA-III
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: The Third Xiangya Hospital of Central South University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Peking University First Hospital (Other); Shanghai Jiao Tong University School of Medicine (Other); Shandong Cancer Hospital and Institute (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Tianjin First Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMU-CIH-IR-004
Record Dates: First submitted 2015-11-03; First posted 2015-11-16 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2015-11

CONDITIONS: Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral bicalutamide once daily on days 1-28. Patients also receive luteinizing-hormone releasing-hormone (LHRH) agonist treatment intramuscularly (IM) on day 8. Treatment with LHRH agonist repeats every 12 weeks for 24 weeks.
  Patients receive cryoablation therapy.
  Interventions: Procedure: Cryoablation therapy; Drug: bicalutamide; Drug: luteinizing-hormone releasing-hormone (LHRH) agonist
- Arm II (Experimental): Patients receive androgen ablation as in arm I. Patients receive external beam radiation therapy.
  Interventions: Radiation: External beam radiation therapy; Drug: bicalutamide; Drug: luteinizing-hormone releasing-hormone (LHRH) agonist

INTERVENTIONS:
Procedure: Cryoablation therapy — Cryoablation therapy
  Arms: Arm I
Radiation: External beam radiation therapy — External beam radiation therapy
  Arms: Arm II
Drug: bicalutamide — bicalutamide
Drug: luteinizing-hormone releasing-hormone (LHRH) agonist — luteinizing-hormone releasing-hormone (LHRH) agonist

SUMMARY:
This trial is going to evaluate tumor control and quality of life in patients with prostate cancer treated with radiotherapy or cryoablation.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the tumor control in patients with prostate cancer treated with radiotherapy or cryoablation
* To determine the quality of life of these patients. OUTLINE: This is a multicenter study. Patients are stratified according to Gleason score (≥ 8 vs 7 vs ≤ 6), persistent prostatic specific antigen (PSA) at allocation (> 0.5 ng/mL vs ≤ 0.5 ng/mL), participating center. Patient are allocated to two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Prostate adenocarcinoma, T3aN0M0, T3bN0M0
* Previously untreated disease or undergone endocrine therapy without reaching to castration resistant prostate cancer
* Survival ≥ 12 months
* WHO performance status 0-2
* white blood cell ≥ 3.5 ×10*9/L
* Platelets ≥ 5×10*9/L
* Hemoglobin ≥ 10 g/dL

Exclusion Criteria:

* History of malignant disease
* History of coronary artery disease
* Uncontrolled infection
* Other concurrent severe or uncontrolled medical disease that could compromise participation in the study (i.e., uncontrolled diabetes mellitus, uncontrolled cardiac disease, uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within the past six months, chronic liver or renal disease, and active upper gastrointestinal tract ulceration)
* Psychological, familial, sociological, or geographical condition potentially hampering compliance with the study treatment and follow-up schedule

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Median PSA progression-free survival in patients responding to the study treatments | Within 12 months after treatment
Quality of Life impact of treatments' side effects measured by change in EORTC QOL-C30 from baseline to 3, 6 and 12 months after treatment | 3, 6 and 12 months after treatment
  European Organization for Research and Treatment of Cancer(EORTC)

SECONDARY OUTCOMES:
Overall survival | 5 year
Disease Specific Survival | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Guo, PhD, Principal Investigator — Tianjin Medical University Cancer Institue and Hospital
Locations (1):
- Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No